CLINICAL TRIAL: NCT03206502
Title: Characterizing Sleep, Stress, and Seizures in Daily Life: An Internet-based Study With the Empatica Embrace Watch and Smartphone-based Diary-alert System
Brief Title: Embrace: Seizure Characterization
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Empatica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-001
Record Dates: First submitted 2016-11-21; First posted 2017-07-02 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Embrace+Alert App (Experimental): Participants are allowed to enter the trial (to use Embrace+Alert app) whether or not they have epilepsy. People without epilepsy may use Alert in this trial even though they are not expected to have seizures, as long as they are willing to mark false positives. Since many people with epilepsy live active lives and appear perfectly healthy outwardly, it is important that their active lifestyle data not trigger false alarms. Allowing healthy participants without epilepsy to contribute active lifestyle data helps us make the detection algorithm even stronger and better.
  Interventions: Device: Embrace + Alert App

INTERVENTIONS:
Device: Embrace + Alert App — Participants will wear an Embrace smartwatch to collect data, and will provide survey/diary information on the occurrence of seizures. The device sends data to the Alert app, which issues either true detections or false alarms when it detects a possible convulsive seizure. Participants are asked to either cancel (in real time) or mark (at a later time) all false alarms using the Alert app.

SUMMARY:
The study is intended to characterize sleep, stress, and seizures in daily life with the Empatica Embrace watch and smartphone-based diary-alert system. The primary study objective is to collect and validate biometric signals from epilepsy patients using the Empatica Embrace watch and compare them to ictal events captured from human (patient and caregiver) reports.

DETAILED DESCRIPTION:
Patients use the Embrace sensor with a smartphone app, "Alert". The sensor attempts to capture convulsive seizure events such as generalized tonic-clonic seizures (GTCS's), and to initiate an alert when such an event is captured. Patients can also enter seizures (captured or not, GTCS or not) into the "Mate" diary, and they can cancel or mark false alarms if Embrace triggered a false alarm.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 1-99
* Anyone (healthy or not) can participate
* Adult participant must either be able to give consent or must have an acceptable surrogate capable of giving consent on their behalf.
* Participants under age 18 must have an adult guardian give informed consent, and if capable, the patient must give informed assent.
* Participants with GTCS must have a functioning smartphone (iOS or Android) that can be paired with the Embrace over a Bluetooth Low Energy connection and agree that it can be kept on or near their person.
* Participants with GTCS (or their surrogate) must be able to identify one or more "designated frequent caregivers," who has a functioning phone, agrees to keep it regularly charged, agrees to receive alerts, and agrees to respond to alerts promptly to the best of their ability.
* Participants must be fluent in the language of the consent forms (Currently limited to English but Spanish and other languages are planned).
* Participants must reside in the United States.

Exclusion Criteria:

* Participants must not have broken or injured skin at the wrist or leg location where Embrace is worn, and they must be able to tolerate wearing Embrace snugly for long periods of time. Thus, they should not have allergies to the material composition of the Embrace watch, or discomfort wearing a wristwatch or leg-band device.
* Participants should not be homeless.
* Participants should not have active dependence on substances that are not currently prescribed by their doctor (e.g. alcohol, pain medications, illegal drugs) or be taking substances that they are not willing to disclose as a study participant.
* Participants must not be pregnant or planning to become pregnant within six months at the time of screening.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the GTCS detection of the Embrace + Alert app | The primary outcome is assessed continuously over the trial period (each new seizure is counted and summed for each person; the average time period is 6 months)
  The number of GTCS automatically detected by Embrace will be compared to the total recorded by the wearer+caregiver in a seizure diary. This fraction is the sensitivity.

SECONDARY OUTCOMES:
False alarm rate of the GTCS detection of the Embrace + Alert app | The secondary outcome is assessed continuously over the trial period (each false alarm is counted and summed for a running total within each person; the average time period is 6 months)
  The number of alerts elicited by Embrace+Alert app that do NOT correspond to convulsive seizures marked in the seizure diary are "false alarms". False alarms can also be explicitly marked by patients.

OTHER OUTCOMES:
System Usability | After one month of use.
  The System Usability Scale will be given to assess system usability

IPD SHARING:
Plan to Share IPD: No